CLINICAL TRIAL: NCT03134131
Title: Expanded Access to ONC201 for Patients With H3 K27M-mutant and/or Midline High Grade Gliomas
Status: No longer available | Type: Expanded Access
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ONC018
Record Dates: First submitted 2017-04-20; First posted 2017-04-28 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2020-10

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — TIC10 compound

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: ONC201 — ONC201 is an oral, small molecule selective antagonist of DRD2 that induces tumor cell death.

SUMMARY:
The objective of this expanded access program is to provide ONC201 to eligible patients with previously-treated glioma that exhibits the H3 K27M mutation and/or that is located in the midline region of the brain.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have one type of diagnosis below:

   1. A glioma that is positive for the H3 K27M mutation (performed in a laboratory with CLIA certification);
   2. A grade III or IV glioma involving the thalamus, hypothalamus, brainstem, cerebellum, midbrain, or spinal cord;
   3. Diffuse intrinsic pontine glioma (DIPG), defined as tumors with a pontine epicenter and diffuse involvement of the pons. These patients are eligible with or without a tissue biopsy.
2. Unequivocal evidence of progressive disease on as defined by RANO criteria or have documented recurrent glioma on diagnostic biopsy.
3. Patient must have had previous therapy that includes radiotherapy.
4. Interval of at least 90 days from the completion of radiotherapy to the first dose of ONC201. If patients are within 90 days of radiotherapy, they may still be eligible if they meet one or more of the following criteria.

   1. Progressive tumor is outside the original high-dose radiotherapy target volume as determined by the treating investigator, or
   2. Histologic confirmation of tumor through biopsy or resection, or
   3. Nuclear medicine imaging, MR spectroscopy, or MR perfusion imaging consistent with true progressive disease, rather than pseudoprogression or radiation necrosis obtained within 28 days of registration.
5. Patient must be at least 3 years of age.
6. Patient must weigh at least 10kg.
7. Patient must be able to swallow and retain orally administered medication. For patients unable to swallow capsules, oral ONC201 will be administered as a liquid formulation in Ora-Sweet.
8. From the projected start of scheduled study treatment, the following time periods must have elapsed from prior anti-cancer treatments: 5 half-lives from any investigational agent, 4 weeks from cytotoxic therapy (except 23 days for temozolomide and 6 weeks from nitrosoureas), 6 weeks from anti-cancer antibodies (except 21 days for bevacizumab), or 4 weeks (or 5 half-lives, whichever is shorter) from other anti-tumor therapies.
9. Contrast-enhanced head CT or brain MRI within 21 days prior to start of study drug.
10. Adequate organ and marrow function as defined below:

    1. Absolute neutrophil count ≥1,000/mm3 without growth factor use ≤ 7 days prior to treatment (cycle 1 day 1, C1D1)
    2. Hemoglobin >8.0 mg/dL without red blood cell transfusion ≤ 3 days prior to C1D1
    3. Total serum bilirubin <1.5 X upper limit of normal (ULN)
    4. AST (SGOT)/ALT (SGPT) ≤2 X ULN; ≤ 5 X ULN if there is liver involvement secondary to tumor
    5. Serum creatinine ≤ 1.5 X ULN (OR creatinine clearance ≥ 60 mL/min/1.73 m2)
11. For patients post pubertal: Female patients must agree to use effective contraception while taking ONC201 and for at least 90 days after completion of treatment. Male patients must be surgically sterile or must agree to use effective contraception while taking ONC201 and for at least 90 days after completion of treatment. The decision of effective contraception will be based on the judgment of the principal investigator.
12. Ability to understand a written informed consent document, and the willingness to sign it. Assent will be obtained when appropriate based on the subjects age.

Exclusion Criteria:

1. Qualifies for participation in an ongoing ONC201 clinical trial or is already participating in an ONC201 clinical trial.
2. Current or planned participation in a study of an investigational agent or using an investigational device.
3. Evidence of diffuse leptomeningeal disease or CSF dissemination.
4. Any known systemic infection that, in the opinion of the investigator, could compromise the safety of the patient, while taking ONC201.

Min Age: 3 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Oncoceutics, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Arrillaga-Romany I, Gardner SL, Odia Y, Aguilera D, Allen JE, Batchelor T, Butowski N, Chen C, Cloughesy T, Cluster A, de Groot J, Dixit KS, Graber JJ, Haggiagi AM, Harrison RA, Kheradpour A, Kilburn LB, Kurz SC, Lu G, MacDonald TJ, Mehta M, Melemed AS, Nghiemphu PL, Ramage SC, Shonka N, Sumrall A, Tarapore RS, Taylor L, Umemura Y, Wen PY. ONC201 (Dordaviprone) in Recurrent H3 K27M-Mutant Diffuse Midline Glioma. J Clin Oncol. 2024 May 1;42(13):1542-1552. doi: 10.1200/JCO.23.01134. Epub 2024 Feb 9. PMID 38335473